CLINICAL TRIAL: NCT06033612
Title: A Randomised, Double Blinded, Placebo-controlled Single and Multiple Ascending Dose Study of Orally Administered RV299 to Evaluate Safety, Tolerability, Pharmacokinetics and Food Effect in Healthy Adult Participants
Brief Title: Safety, Tolerability, Pharmacokinetics, and Food Effect Study of RV299 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVD001; C5251001 (Other: Alias Study Number)
Record Dates: First submitted 2022-08-11; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; bronchiolitis; lower respiratory tract infection; LRTI
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A and B (Cohorts 1 -2) participants and care providers will remain blinded to study allocation. Part B (Cohort 3) and Part C participants will not be blinded to their study treatment.
  The placebo bottle will be covered with a paper sleeve to ensure contents remain blinded. Pharmacy staff preparing investigational products will not be blinded to drug assignment. During the trial, individual randomisation codes will be kept in the site's clinical trials pharmacy, accessible to the pharmacy personnel only. Drug accountability will be reviewed by an unblinded CRA.
  Sponsor staff involved in clinical decision-making (e.g. Safety Review Committee) will be blinded to drug assignment. Sponsor staff performing PK analysis will be unblinded but will deliver blinded PK data and reports to the blinded sponsor and Investigator teams. A cardiologist will examine all ECG recordings of Part B participants with readers blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A Single Ascending Dose (SAD) - RV299/Placebo (Experimental): Participants will receive RV299 or placebo as a single dose on Day 1. Sentinel dosing will be used (one on RV299 and one on placebo) before the rest of the cohort are dosed together.
  Interventions: Drug: RV299; Drug: Placebo
- Part B Multiple Ascending Dose (MAD) - RV299/Placebo (Experimental): Participants will receive RV299 or placebo twice daily on Day 1-4 and a single dose on Day 5. Participants in each cohort will receive ascending doses of RV299, depending on emerging safety and PK data.
  Part B, Cohort 3 will investigate interaction between midazolam and RV299. Participants will receive a single dose of midazolam on Day 1 and Day 7, and receive RV299 twice daily on Days 2 - 6
  Interventions: Drug: RV299; Drug: Placebo; Drug: Midazolam
- Part C Food Effect (FE)- RV299 (Experimental): Participants will receive RV299 as a single dose on Day 1 and Day 5; treatment will be administered in the first treatment period fasted and the second treatment period fed (or vice versa).
  Interventions: Drug: RV299

INTERVENTIONS:
Drug: RV299 — Oral Suspension
Drug: Placebo — matching placebo
  Arms: Part A Single Ascending Dose (SAD) - RV299/Placebo; Part B Multiple Ascending Dose (MAD) - RV299/Placebo
Drug: Midazolam — pre-filled oral syringe
  Arms: Part B Multiple Ascending Dose (MAD) - RV299/Placebo

SUMMARY:
The main aims of the study are to assess the safety, tolerability, pharmacokinetics and food effects of RV299 compared to Placebo in healthy adult participants.

The study consists of three parts: single ascending dose (Part A), multiple ascending doses (Part B) and food effect (Part C) in Caucasian participants.

DETAILED DESCRIPTION:
This is a randomised, double blind, placebo-controlled Phase I study to assess the safety, tolerability, pharmacokinetics and food effect of RV299 in healthy participants aged ≥ 20 to ≤ 40 years.

The clinical study consists of 3 parts (Parts A - C):

Part A: single ascending doses (SAD) of RV299 in healthy adult Caucasian participants (up to 3 dose levels of RV299 in 3 cohorts; 6 participants/cohort)

Part B: multiple ascending doses (MAD) of RV299 in healthy adult Caucasian participants (up to 2 dose levels of RV299 in 2 cohorts of 8 participants dosed for 5 consecutive days). Part B will incorporate a drug-drug interaction (DDI) design to investigate interaction between RV299 and midazolam in one cohort (Cohort 3) of 8 participants.

Part C: food effect (FE) in healthy adult Caucasian participants (one cohort of 8 participants to be randomised to receive either RV299 in the first treatment period fasted and in the second treatment period fed, or vice versa)

The study will be conducted as an adaptive integrated design since various study parts can be triggered at appropriate times during the conduct of other parts of the study. Dose escalation to the following scheduled dose or progression to a consecutive part of the study will only occur after satisfactory review of all safety, tolerability and pharmacokinetic (PK) data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, Caucasian, aged greater than or equal to 20 to less than or equal to 40 years at the date of signing informed consent.
2. Participants in Caucasian cohorts should be distinguished by very light to brown skin pigmentation and straight to wavy or curly hair, and should be indigenous to Europe, northern Africa, western Asia, India. This includes Caucasian participants from North America, Australia and South Africa.
3. Healthy as defined by: a) the absence of clinically significant illness and surgery within four weeks prior to dosing; b) the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
4. Participants must agree to use contraceptive requirements as described in the study protocol for the applicable duration.
5. Participants must agree not to donate sperm or ova from the time of the first administration of trial medication until 3 months after three months after the last follow-up visit.
6. Participants must have a body mass index (BMI) between 18.0-25.0 kg/m² inclusive at screening.
7. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation that is reasonably likely to interfere with the participant's participation in or ability to complete the trial as assessed by the Investigator.
8. Ability to provide written, personally signed, and dated informed consent.
9. An understanding, ability, and willingness to fully comply with trial procedures and restrictions.

Exclusion Criteria:

1. Current or recurrent disease (e.g., cardiovascular, haematological, neurological, endocrine, immunological, renal, hepatic or gastrointestinal or other conditions) that could affect the action, absorption, or disposition of RV299, or could affect clinical assessments or clinical laboratory evaluations.
2. Current or relevant history of physical or psychiatric illness that are not stable or may require a change in treatment, use of prohibited therapies during the trial or make the participant unlikely to fully comply with the requirements of the trial or complete the trial, or any condition that presents undue risk from the investigational product or trial procedures.
3. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial may influence the result of the trial, or the participant's ability to participate in the trial.
4. Use or intention to use any medications/products that are known inhibitors of the CYP3A4 enzymes or substrates of Aldehyde oxidase (AO), Pglycoprotein (PgP) or Breast Cancer Resistance Protein (BCRP) for 2 weeks prior to Day 1 of the dosing period up to the follow-up visit. (The Indiana University (2016) "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors of CYP3A) (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
5. The history or presence of any of the following cardiac conditions known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.
6. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes. (Participants with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.)
7. Has vital signs outside of the following normal range at screening or Day -1/Day-2.
8. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening;
9. Has a haemoglobin, platelet count, total white blood cell count, lymphocyte or monocyte count less than lower limit of normal (LLN) (up to two repeats may be taken).
10. Has total bilirubin, ALT or AST consistently greater than ULN at Screening (up to two repeats may be taken).
11. Any other abnormal findings on vital signs, ECG, physical examination or laboratory evaluation of blood and urine samples that the Investigator judges as likely to interfere with the trial or pose an additional risk in participating.
12. Positive test results for alcohol or drugs of abuse at screening or Day-1/Day-2.
13. History or clinical evidence of substance and/or alcohol abuse within the 2 years before screening.
14. Treatment with an investigational drug within 90 days or 5 half-lives preceding the first dose of trial medication (or as determined by the local requirement, whichever is longer).
15. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine containing products in any form (e.g., gum, patch, electronic cigarettes) within 3 months prior to the planned first day of dosing.
16. Has used any other prescription medication within 14 days or 10 half-lives (whichever is longer) prior to Day 1 of the dosing period that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating.
17. Has used any over-the-counter medication (including multivitamin, herbal, or homeopathic preparations; excluding paracetamol - up to 2g paracetamol per day permitted) during the 7 days or 10 half-lives of the drug (whichever is longer) prior to Day 1 of the dosing period, that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating.
18. Consumption of herbal remedies or dietary supplements containing St. John's Wort in the three weeks before the planned Day 1 of the dosing period.
19. Known or suspected intolerance or hypersensitivity to the investigational product, any closely related compound, or any of the stated ingredients.
20. History of significant allergic reaction (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).
21. Donation of blood or blood products (excluding plasma) within 90 days prior to trial medication administration.
22. Has a mental incapacity or language barriers precluding adequate understanding, co-operation, and compliance with the trial requirements.
23. An inability to follow a standardised diet and meal schedule or inability to fast, as required during the trial.
24. Participants with veins on either arm that are unsuitable for intravenous puncture or cannulation.
25. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), randomisation, participation, or enrolment in this trial. Participants who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved.
26. Participants who have received or are planning on receiving a COVID-19 vaccination two weeks before first dose administration, or within one week after the final follow-up visit for the study.
27. Known or suspected intolerance or hypersensitivity to the investigational product, the non-investigational product (midazolam), any closely related compound, or any of the stated ingredients.
28. Female participants currently on combined hormonal contraception or hormonal replacement therapy containing oestradiol or ethinyloestradiol.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAE) as assessed by CTCAE V5.0. | Part A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Listings and summary tables of AEs will be based on TEAEs (defined as events starting, or worsening, after the first dose of RV299).
Evaluate the proportion of participants with clinically significant shifts in haematology/clinical chemistry/coagulation/urinalysis values from baseline following dosing with RV299 | Part A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Blood and urine tests will be conducted at a central laboratory. Results at each visit will be summarized using the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate the proportion of subjects with changes in ECG measurements from baseline following dosing with RV299 | Part A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Parameters collected will be:
  PR interval (msec); QRS interval (msec); QT interval (msec); QTcB interval (msec); QTcF interval (msec); Heart rate (bpm). Results at each visit will be summarized using the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV299 by assessing changes from baseline in tympanic temperature (vital sign parameters) | Part A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Tympanic temperature will be collected in degrees Celsius (°C). Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV299 by assessing changes from baseline in blood pressure (BP) (vital sign parameters). | Part A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Blood pressure (systolic and diastolic) will be measure in mm Hg. Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV299 by assessing changes from baseline in heart rate (HR) (vital sign parameters). | PPart A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Heart rate will be measure in beats per minute (bpm). Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV299 by assessing changes from baseline in respiratory rate (vital sign parameters). | Part A: 7 days after single dose; Part B: 28 days after final dose; Part C: 7 days after final dose
  Respiratory rate will be measured in breaths per minute. Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Assess area under the plasma concentration versus time curve (AUC) of midazolam (as index substrate) from 0 to 24 hours post-dose (AUC0-24h) before and after dosing with RV299. | Part B Cohort 3 only: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 13, 16, and 24 hours following administration of midazolam on Day 1 and Day 7.
  Pharmacokinetic analysis will include listings and summaries of midazolam concentration by time point and analysis of relationship with dose and body weight.
Assess time to maximum plasma concentration (tmax) of midazolam (as index substrate) before and after dosing with RV299. | Part B Cohort 3 only: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 13, 16, and 24 hours following administration of midazolam on Day 1 and Day 7.
  Pharmacokinetic analysis will include listings and summaries of midazolam concentration by time point and analysis of relationship with dose and body weight
Assess terminal half life of (t1/2) of midazolam (as index substrate) before and after dosing with RV299. | Part B Cohort 3 only: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 13, 16, and 24 hours following administration of midazolam on Day 1 and Day 7.
  Pharmacokinetic analysis will include listings and summaries of midazolam concentration by time point and analysis of relationship with dose and body weight
Assess maximum plasma concentration (Cmax) of midazolam (as index substrate) before and after dosing with RV299. | Part B Cohort 3 only: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 13, 16, and 24 hours following administration of midazolam on Day 1 and Day 7.
  Pharmacokinetic analysis will include listings and summaries of midazolam concentration by time point and analysis of relationship with dose and body weight

SECONDARY OUTCOMES:
Characterise plasma pharmacokinetics (PK) of RV299 by assessing time to maximum plasma concentration (tmax) following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess terminal half-life (t1/2) of RV299 following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess rate constant (λz) of RV299 following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess maximum plasma concentration (Cmax) of RV299 following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess area under the plasma concentration versus time curve (AUC) of RV299 from time zero to last quantifiable plasma concentration (AUC0-t) following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess area under the plasma concentration versus time curve (AUC) from time zero to 24 hours post-dose (AUC0-24h) following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 24 hours after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess area under the plasma concentration-time curve of RV299 from time zero to infinity (AUC0-inf) following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess accumulation ratio of RV299 based on AUC0-tau following multiple doses of RV299. | Part B only: pre-dose (Day 1) to 7 days after final dose of RV299 (at Day 5)
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess minimum blood plasma concentration (Cmin) of RV299 between administration of two doses of RV299. | Parts B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess plasma clearance (rate of removal of RV299 from plasma) (CL/F) following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess apparent volume of distribution (VZ/F) of RV299 following single and multiple doses of RV299. | Parts A, B and C: pre-dose (Day 1) to 7 days after final dose of RV299
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess area under the plasma concentration versus time curve (AUC) of RV299 after dosing in the fed and fasted states. | Part C only: pre-dose (Day 1) to 7 days after second (final) dose (Day 5).
  First dose of RV299 will be given while participant is in the fasted state; second dose will be given after patient has eaten (and vice-versa). Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight.
Assess maximum plasma concentration (Cmax) of RV299 after dosing in the fed and fasted states. | Part C only: pre-dose (Day 1) to 7 days after second (final) dose (at Day 5).
  First dose of RV299 will be given while participant is in the fasted state; second dose will be given after patient has eaten (and vice-versa). Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight.
Characterise steady-state plasma pharmacokinetics (PK) of RV299 following multiple doses of RV299 by comparing AUC against dosing intervals. | Part B only: pre-dose (Day 1) to 7 days after final dose of RV299 (at Day 5).
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight
Assess area under the plasma concentration versus time curve from time zero to 12 hours post-dose (AUC0-12) following multiple doses of RV299. | Part B only: pre-dose to 12 hours following administration of first dose of RV299 (Day 1) and final dose (Day 5)
  Pharmacokinetic analysis will include listings and summaries of RV299 concentration by time point, derived PK, parameters and analysis of relationship with dose and body weight

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Richmond Pharmacology Ltd, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=REVD001